CLINICAL TRIAL: NCT01383408
Title: Distinction Between Lung Cancer and Gynecological Cancers by Exhalation Analysis and Canine Scent Detection
Brief Title: Distinction Between Lung Cancer and Gynecological Cancers by Canine Scent Detection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inconsistent training status of sniffer dogs
Sponsor: Schillerhoehe Hospital (Other)
Collaborators: Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other)
Responsible Party: Principal Investigator, Thorsten Walles, Principal Investigator, Schillerhoehe Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: KSH-TCH-IIT-2011-1
Record Dates: First submitted 2011-06-24; First posted 2011-06-28 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Lung Cancer; Breast Cancer; Ovarian Cancer
Keywords: breath sample analysis; exhalation analysis; volatile organic compounds; screening; lung cancer; breast cancer; ovarian cancer; canine scent detection
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- healthy individual (Sham Comparator): healthy individual with no lung disease and no history of cancer including lung cancer
  Interventions: Other: exhalation analysis of breath sample
- lung cancer (Experimental): patients with histologically confirmed lung cancer, but no history of other cancer
  Interventions: Other: exhalation analysis of breath sample
- breast cancer (Experimental): patients with histologically confirmed breast cancer, but no history of other cancer
  Interventions: Other: exhalation analysis of breath sample
- ovarian cancer (Experimental): patients with histologically confirmed ovarian cancer, but no history of other cancer
  Interventions: Other: exhalation analysis of breath sample

INTERVENTIONS:
Other: exhalation analysis of breath sample — study participants exhale 5 times into a test tube; test tube is presented to sniffer dogs for analysis

SUMMARY:
Previous studies have shown that specially trained sniffer dogs are capable to discriminate breath samples of patients with lung cancer and healthy individuals. So far it is not known whether this differentiation is specific for lung cancer or just identifies any form of (solid) tumor. Therefore, the dog's ability to differentiate between lung cancer, breast cancer and ovarian cancer is tested.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed lung or breast or ovarian cancer

Exclusion Criteria:

* other cancers
* previous medical intervention within the last 14 days before gathering of the breath sample

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 752 (Actual)
Dates: Start 2011-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Specificity for Lung Cancer | breath samples will be tested within 40 days after gathering
  exhalation analysis by sniffer dogs is able to differentiate breath samples of patients with lung cancer from those of patients with other (tested) cancers

SECONDARY OUTCOMES:
Discriminability of breast and ovarian cancer | breath samples will be tested within 40 days after gathering
  exhalation analysis by sniffer dogs is able to differentiate breath samples of patients with breast cancer from those of patients with other ovarian cancer

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Walles, MD, Principal Investigator — Schillerhoehe Hospital; Godehard Friedel, MD, Study Chair — Schillerhoehe Hospital; Wolfgang Simon, MD, Study Chair — Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF)
Locations (2):
- Germany (2):
  - Schillerhoehe Hospital, Gerlingen, Baden-Wurttemberg
  - Robert Bosch Hospital, Stuttgart, Baden-Wurttemberg

REFERENCES:
- [Background] Boedeker E, Friedel G, Walles T. Sniffer dogs as part of a bimodal bionic research approach to develop a lung cancer screening. Interact Cardiovasc Thorac Surg. 2012 May;14(5):511-5. doi: 10.1093/icvts/ivr070. Epub 2012 Feb 17. PMID 22345057
- [Background] Ehmann R, Boedeker E, Friedrich U, Sagert J, Dippon J, Friedel G, Walles T. Canine scent detection in the diagnosis of lung cancer: revisiting a puzzling phenomenon. Eur Respir J. 2012 Mar;39(3):669-76. doi: 10.1183/09031936.00051711. Epub 2011 Aug 18. PMID 21852337